CLINICAL TRIAL: NCT02375295
Title: A Prospective Randomized Trial of 2 Weeks vs 3 Months of Antibiotics Post Percutaneous Nephrolithotomy for the Prevention of Infection-Related Kidney Stones
Brief Title: Struvite Stones Antibiotic Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H13-02514
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Kidney Stones
Keywords: struvite; infection; stones; calculi; antibiotics
MeSH Terms: conditions — Kidney Calculi; Infections; Calculi | interventions — Ciprofloxacin; Nitrofurantoin; Cephalexin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: 2 weeks Abx post PCNL (Experimental): Oral antibiotics: ciprofloxacin, cotrimoxazole-trimethoprim, or macrodantin are administered for 2 weeks at full dose.
  Interventions: Drug: ciprofloxacin, cotrimoxazole-trimethoprim, macrodantin
- Arm B: 12 weeks/3 months Abx post PCNL (Active Comparator): Oral antibiotics: ciprofloxacin, cotrimoxazole-trimethoprim, or macrodantin are administered for 2 weeks at full dose followed by a suppressive dose for another 10 weeks (total = 12 weeks or 3 months).
  Interventions: Drug: ciprofloxacin, cotrimoxazole-trimethoprim, macrodantin

INTERVENTIONS:
Drug: ciprofloxacin, cotrimoxazole-trimethoprim, macrodantin — Approved antibiotics used routinely will be given at the physician's discretion with the patient: ciprofloxacin, cotrimoxazole-trimethoprim, or macrodantin
  Other Names: Keflex, Macrobid, co-trimoxazole

SUMMARY:
The aim of this research is to determine an effective antibiotic regimen following definitive surgical therapy of kidney stones caused by bacterial infection (struvite stones).

DETAILED DESCRIPTION:
Struvite stones or infection stones are a subset of kidney stones that are related to bacterial infection. They only make up 15% of all kidney stones, but account for a much higher percentage of mortality (up to 67%) compared to other stones-due to the infectious component. Treatment is to ensure 100% eradication of the stone with surgery followed by antibiotics to eliminate the infection. Failure to eliminate the bacteria results in the stone growing back quickly. It is unknown how long antibiotics should be administered immediately after surgery-some urologists give 2-4 weeks while others give 2-3 months. We seek to randomize patients to receive 2 weeks of antibiotics or 3 months of antibiotics after surgery to remove all the kidney stones. We will see patients at 3, 6, and 12 months with x-rays and to test their urine for bacterial infections. This is a multi-centre study with participating 12 sites across North America.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female.
2. No age restriction.
3. Diagnosed with an infection related stone.
4. Medically fit for definitive surgical management of stone.
5. Life expectancy greater than one year.
6. Stone free after definitive surgical therapy defined as fragments less than 3mm.

Exclusion Criteria:

1. Patients with medical comorbidities preventing them from definitive surgical therapy.
2. Patients with persistent stone burden following definitive surgical therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2015-03; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
any recurrent kidney stones | 6 months
  Radiologic recurrence of calculi in the location of original treatment at or before 6 months following definitive surgical therapy.

SECONDARY OUTCOMES:
UTI | 1 year
  Positive urine cultures at any point within 1 year from surgical therapy.
treated site stone recurrence rates | 1 year
  Radiologic recurrence of calculi in the location of original treatment at or before 12 months following definitive surgical therapy
Clostridiuum difficile colitis | 1 year
  Antibiotic related complications such as Clostridiuum difficile colitis infections.
ER visit | POD1
  In hospital sepsis and febrile episodes.
Readmission for sepsis. | 3 months
  Readmission for sepsis.
Readmission for renal colic | 3 months
  Readmission for renal colic
Morbidity or mortality related to sepsis or renal failure | 3 months
  Morbidity or mortality related to sepsis or renal failure
Repeat surgical procedures for stone recurrence | 3 months
  Repeat surgical procedures for stone recurrence
Ancillary procedures for stones such as ureteric stenting and nephrostomy tubes | 3 months
  Ancillary procedures for stones such as ureteric stenting and nephrostomy tubes

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia
Locations (12):
- United States (11):
  - Mayo Clinic - Scottsdale/Phoenix, AZ, Scottsdale, Arizona
  - University California San Diego, San Diego, California
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, MN, Rochester, Minnesota
  - Dartmouth University, Lebanon, New Hampshire
  - New York University, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Athens, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
- The Stone Centre, VGH/UBC, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No